CLINICAL TRIAL: NCT02646670
Title: Efficacy of Ranibizumab Therapy With Aflibercept in Patients With Diabetic Macular Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARVO R2 2016
Record Dates: First submitted 2015-12-02; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Retinal Diseases
Keywords: diabetic macular edema; aflibercept; ranibizumab
MeSH Terms: conditions — Retinal Diseases | interventions — Ranibizumab; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ranibizumab (Active Comparator): - In the first group will be held three applications of intravitreal ranibizumab 0.1 ml . This group will be five about patients about any age, with diabetic macular edema randomly chosen
  Interventions: Drug: Ranibizumab
- Aflibercept (Active Comparator): - In the second group will be held three applications of Intravitreal Aflibercept 0.1 ml. This group will be about five patients about any age, with diabetic macular edema randomly chosen
  Interventions: Drug: Aflibercept
- Ranibizumab and Aflibercept (Active Comparator): - In this group will be held two applications of 0.1 ml Aflibercept(the first and the third doses) interspersed with one application of Ranibizumab 0.1 ml(the second dose). This group will be about five patients about any age, with diabetic macular edema randomly chosen
  Interventions: Drug: Ranibizumab and Aflibercept
- Aflibercept and Ranibizumab (Active Comparator): - This group will be held two applications of Ranibizumab 0.1 ml(the first and the third doses) interspersed with one application of Aflibercept 0.1 ml(the second dose). This group will be five about patients about any age, with diabetic macular edema randomly chosen
  Interventions: Drug: Aflibercept and ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — - In the first group will be held three applications of intravitreal ranibizumab 0.1 ml, with one application every month and follow up with Optical Coherence Tomography
  Arms: Ranibizumab
Drug: Aflibercept — - In the second group will be held three applications of Intravitreal Aflibercept 0.1 ml, with one application each month followed by monitoring with Optical Coherence Tomography
  Arms: Aflibercept
Drug: Ranibizumab and Aflibercept — - The third group will be held two applications of Ranibizumab 0.1 ml interspersed with one application of Aflibercept 0.1 ml in the second month and subsequent evaluation with Optical Coherence Tomography
  Arms: Ranibizumab and Aflibercept
Drug: Aflibercept and ranibizumab — - In the fourth group will be held two applications of 0.1 ml Aflibercept interspersed with one application of Ranibizumab 0.1 ml in the second month and subsequent evaluation with Optical Coherence Tomography
  Arms: Aflibercept and Ranibizumab

SUMMARY:
The purpose of this study in to compare the efficacy of treatment of diabetic macular edema (DME) using Ranibizumab (Lucenti®), Aflibercept (Eylea®) and Aflibercept (Eylea®) plus Ranibizumab (Lucentis®).

It is a randomized clinical trial that will evaluate the efficacy of the combination of two substances currently used in the treatment of DME. Will be allocated in different four groups randomly pacients who receive treatment with intravitreal injections of ranibizumab, aflibercept or a combination of aflibercept and ranibizumab.

DETAILED DESCRIPTION:
Interventions will be carried out with intravitreal injections in patients with formal indications of diabetic macular edema treatment previously assessed with complete eye examination in Goiania Eye Institute(Instituto de Olhos de Goiânia)

Patients will be divided into four groups:

* In the first group will be held three applications of intravitreal ranibizumab 0.1 ml, with one application every month and follow up with Optical Coherence Tomography on days 1, 3, 5, 10 and 30 following the application.
* In the second group will be held three applications of Intravitreal Aflibercept 0.1 ml, with one application each month followed by monitoring with Optical Coherence Tomography on days 1, 3, 5, 10 and 30 subsequent
* The third group will be held two applications of Ranibizumab 0.1 ml interspersed with one application of Aflibercept 0.1 ml in the second month and subsequent evaluation with Optical Coherence Tomography on days 1, 3, 5, 10 and 30.
* In the fourth group will be held two applications of 0.1 ml Aflibercept interspersed with one application of Ranibizumab 0.1 ml in the second month and subsequent evaluation with Optical Coherence Tomography on days 1, 3, 5, 10 and 30.

ELIGIBILITY:
Inclusion Criteria:

* patients with Diabetic macular edema

Exclusion Criteria:

* patients without diabetic macular edema, or with diabetic macular edema with other disease that can make confuse about the diagnose

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of Ranibizumab Therapy with Aflibercept in Patients with Diabetic Macular Edema | 3 months
  Were evaluated the therapy with two different drugs used in diabetic retinopathy, and for this were separated twenty patients in four groups:
  * First group will be held three applications of intravitreal ranibizumab 0.1 ml, and follow up with OCT.
  * Second group will be held three applications of Intravitreal Aflibercept 0.1 ml, and followed by monitoring with OCT.
  * Third group will be held two applications of 0.1 ml Aflibercept interspersed with one application of Ranibizumab 0.1 ml in the second month and subsequent evaluation with OCT.
  * Fourth group will be held two applications of Ranibizumab 0.1 ml interspersed with one application of Aflibercept 0.1 ml in the second month and subsequent evaluation with OCT.
  In all this groups will be observe the time of reduction of macular edema in the days 1, 3, 5, 10 and 30.